CLINICAL TRIAL: NCT01158443
Title: Behavioral Activation/Armodafinil to Treat Fatigue in HIV/AIDS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Responsible Party: Principal Investigator, Judith G. Rabkin, PhD, Research Scientist VI, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R34MH090843 (NIH)
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2014-03

CONDITIONS: Hiv; Fatigue; Goals
Keywords: HIV+; fatigue; return to work
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Fatigue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral activation therapy (Experimental): The Behavioral Activation Program for Energy and Productivity (BA-PEP) is a manualized, 8-session intervention, scheduled to coincide with maintenance armodafinil treatment. It is a structured counseling program with homework, short-term activities and goals, and includes problem-solving, identification of barriers and strategies for their resolution, with an ongoing focus on achieving employment or training.
  Interventions: Behavioral: Behavioral Activation Therapy
- supportive counseling (SC) (Placebo Comparator): Supportive counseling is designed to create an empathic, accepting environment, to direct attention to the patient's feelings and to facilitate acceptance of affective experience using supportive statements, reflective listening and empathic communications.
  Interventions: Behavioral: Supportive Counseling

INTERVENTIONS:
Behavioral: Behavioral Activation Therapy — 8 session, manualized intervention. Homework, short-term activities and goals specified, problem solving skills.
  Other Names: BA
  Arms: Behavioral activation therapy
Behavioral: Supportive Counseling — 8 sessions of manualized supportive counseling. Frequency and duration are designed to match the Behavioral Activation arm.
  Arms: supportive counseling (SC)

SUMMARY:
This is an integrated medication/behavioral intervention program to increase energy, activity level and goal attainment in a sample of HIV+ adults whose presenting problems include both clinically significant fatigue and unmet vocational goals. Based on previous studies, the investigators found that many patients fail to achieve desired goals even though energy is restored by medication. To address this failure of goal attainment, the investigators will evaluate a behavioral intervention, originally based on Behavioral Activation Treatment for Depression, and modified as Behavioral Activation Program for Energy and Productivity or BA-PEP. The intervention will be conducted with patients who experience clinically significant fatigue and who want to work or receive work-related training (paid or volunteer, part time or full time) or education once energy improves with medication (armodafinil).

DETAILED DESCRIPTION:
The investigators propose an integrated medication/behavioral intervention program to increase energy, activity level and goal attainment in a sample of people with HIV/AIDS whose presenting problem is clinically significant fatigue and unmet vocational goals. Based on a recently completed randomized controlled trial (RCT) of modafinil and ongoing RCT of armodafinil, the investigators found that many patients fail to achieve desired goals even though energy is restored by medication. To address this failure of goal attainment, the team will develop and pilot a behavioral intervention, originally based on Behavioral Activation Treatment for Depression of Lejuez et al. and modified by Dr. Daughters as "Behavioral Activation Program for Energy and Productivity, or 'BA-PEP'". The intervention will be conducted with patients who experience significant fatigue, and who want to work or get work-related training or education once their energy improves with armodafinil treatment. It is intended for eventual implementation in HIV clinics and community agencies with work development programs.

The intervention development includes both formative work and pilot studies. The formative work comprises in-depth patient interviews, focus groups with providers, a Project Advisory Board, and a separate Work Group. Their input will be used to modify their BA-PEP intervention to promote achievement of goals selected by each patient, once fatigue has been ameliorated with armodafinil, and to further adapt the attention control supportive counseling intervention.

With this input, the investigators will conduct an exploratory study using BA-PEP with 12 patients responsive to armodafinil. After further modifications, investigators will conduct a feasibility trial with 30 armodafinil-responsive patients randomized 2:1 to BA-PEP or an attention control, supportive counseling. The main behavioral outcome is employment or taking classes (measured by Goal Attainment Scaling methodology). Secondary outcomes are reduced avoidance/increased activation (measured by the Behavioral Activation for Depression Scale), and increased environmental interactions (measured by the EROS: Environmental Rewards Observation Scale). Finally, they will develop training and supervision manuals to guide implementation.

ELIGIBILITY:
Inclusion Criteria:

* HIV+, ages 18-70
* Under the care of a medical provider
* Clinically significant fatigue
* Speaks English
* Able and willing to give informed consent
* Patient seeks either work or vocational training but is blocked from doing so by current fatigue

Exclusion Criteria:

* Primary care provider does not approve of study participation
* Medical rule-outs such as anemia, hypothyroidism, hypogonadism or other condition that may account for fatigue
* Abnormal EKG
* Untreated major depressive disorder; psychosis, bipolar disorder
* Current substance abuse/dependence
* Clinically significant suicidal ideation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-07; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Employment or enrollment in vocational classes as measured by Goal Attainment Scaling | 6 months
  Goal Attainment Scaling assesses degree of success in reaching a pre-specified set of goals initially enumerated at study entry, with a 5-point score range. A score of zero is assigned to success in attaining the specified goal, with 2 greater and 2 lesser levels of accomplishment also specified.

SECONDARY OUTCOMES:
Increased environmental interactions as measured by the EROS: Environmental Rewards Observation Scale. | 6 months
  This is a standardized 10-item scale with a 4-point agree/disagree response format.

CONTACTS AND LOCATIONS:
Overall Officials: Judith G Rabkin, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Rabkin JG, McElhiney MC, Rabkin R, McGrath PJ. Modafinil treatment for fatigue in HIV/AIDS: a randomized placebo-controlled study. J Clin Psychiatry. 2010 Jun;71(6):707-15. doi: 10.4088/JCP.09m05171bro. Epub 2010 May 4. PMID 20492840